CLINICAL TRIAL: NCT03710161
Title: Effect of Vitamin D Supplementation on Balance in Patients With Chronic Kidney Disease
Brief Title: Effect of Vitamin D Supplementation on Balance in CKD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was stopped due to the COVID pandemic
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0608-18-FB
Record Dates: First submitted 2018-10-15; First posted 2018-10-18 (Actual); Results first posted 2021-06-14 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Renal Insufficiency, Chronic; Kidney Failure, Chronic
Keywords: dialysis; end stage renal disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 4000 IU Vitamin D (Experimental): 4000 IU Vitamin D taken daily for six months
  Interventions: Drug: Vitamin D
- 800 IU Vitamin D (Active Comparator): 800 IU Vitamin D taken daily for six months
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — Vitamin D taken in two different dosages daily for six months.
  Other Names: 25(OH)D

SUMMARY:
Patients with end-stage renal disease on dialysis (ESRD5D) are 4-5x more likely to suffer from a fracture. Fractures can occur spontaneously but typically occur after a fall. Further, 70-90% of patients with ESRD5D are vitamin D deficient. Vitamin D supplementation has become routine care for many in this patient population, but evidence is lacking to support this practice. The proposed projects objective is to gather needed preliminary data regarding the effects of vitamin D supplementation on balance and muscle strength in patients with ESRD5D.

DETAILED DESCRIPTION:
In 2009, ~6% of the annual Medicare budget was spent to treat people with end-stage renal disease on dialysis (ESRD5D), making chronic kidney disease (CKD) an important and costly health problem affecting the United States. These patients are 4-5x more likely to suffer from a fracture. Fractures can occur spontaneously but typically occur after a fall. Further, 70-90% of patients with ESRD5D are vitamin D deficient. Vitamin D supplementation has become routine care for many in this patient population; without evidence to support this practice. While studies on the elderly document the effect of vitamin D in decreasing fall risk, findings are inconclusive for those elderly individuals with ESRD5D. The proposed projects objective is to gather needed preliminary data regarding the effects of vitamin D supplementation on balance and muscle strength in patients with ESRD5D. Thirty patients with ESRD5D will be recruited and randomized into two groups: 1) 4000 or 2) 800 IU oral, vitamin D taken daily. Men and women (ages 21-70 years) will be recruited from among patients receiving hemodialysis at a UNMC-directed dialysis facility. Other inclusion criteria include 1) likely to be able to complete the study; 2) ambulatory, without a walking aid; 3) able to complete questionnaires interactively with a research nurse; and 4) greater than 3 months on hemodialysis. Exclusion criteria include patients on peritoneal dialysis, allergy to vitamin D, liver disease, intestinal disorders that would interfere with vitamin D absorption; vitamin D supplements >800 IU per day, glucocorticoids, anticonvulsants, drug therapies for osteoporosis. All patients will be receiving standard of care per their nephrologist. Functional data will be collected at baseline, three, and six months. Data collected will include balance, muscle strength, and falls. Data to monitor vitamin D levels and calcium will be pulled from their medical record. There is no follow up after the six month long study.

ELIGIBILITY:
Inclusion Criteria:

* must be likely to be able to complete the study
* must be able to walk without a walking aid
* must be able to complete questionnaires interactively research staff
* must have been on dialysis for greater than 3 months
* all patients must be receiving standard of care per their nephrologist

Exclusion Criteria:

* peritoneal dialysis
* an allergy to vitamin D
* liver disease
* intestinal disorders that would interfere with vitamin D absorption
* taking vitamin D supplements >800 IU per day, glucocorticoids, anticonvulsants, or other drug therapies for osteoporosis
* are pregnant

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenna Yentes, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska at Omaha, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
De -identified data will be published as supplementary data to manuscripts.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 4000 IU Vitamin D | 800 IU Vitamin D
Started | 3 | 2
Completed | 0 (Study halted due to COVID pandemic) | 0 (Study halted due to COVID pandemic)
Not Completed | 3 | 2
Not completed — Study halted due to COVID pandemic | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 4000 IU Vitamin D | 800 IU Vitamin D | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (5.7) | 48.5 (5.5) | 55.6 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 0 | 1 | 1
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 2 | 5
Height (cm) [Mean (Standard Deviation); unit: cm] | 174.7 (5.0) | 166.5 (2.5) | 171.7 (5.8)
Mass (kg) [Mean (Standard Deviation); unit: kg] | 97.0 (21.5) | 112.3 (22) | 103.1 (22.9)
Resting HR [Mean (Standard Deviation); unit: bpm] | 69.3 (12.3) | 69 (1) | 69.2 (9.5)

OUTCOME MEASURES:

1. Primary Outcome: Timed up and go
Description: This measures fall risk. The measure is a length of time it takes to complete a walking test. A longer score indicates a longer amount of time to complete the test. A shorter amount of time is considered better.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | 4000 IU Vitamin D | 800 IU Vitamin D
Number analyzed (Participants) | 3 | 2
seconds | 11.4 (5.2) | 9.8 (1.7)

2. Primary Outcome: Fullerton Advanced Balance Scale
Description: This 10 item assessment measures one's balance. Scores can range between 0-40. A score of 40 is considered the best performance.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 4000 IU Vitamin D | 800 IU Vitamin D
Number analyzed (Participants) | 3 | 2
score on a scale | 25.3 (6.9) | 34 (5)

3. Primary Outcome: Gait Speed Over 20 Meters
Description: Walking speed is measured over distance of 20 meters. Walking speed is measured in meters per second. A faster walking speed is considered better. Time in seconds needed to cover 20 meters while walking is reported.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: seconds (Time in seconds to walk 20m)
Arm/Group | 4000 IU Vitamin D | 800 IU Vitamin D
Number analyzed (Participants) | 3 | 2
seconds (Time in seconds to walk 20m) | 22.2 (6.6) | 20.0 (.7)

4. Secondary Outcome: Strength of the Quadriceps (Right Leg)
Description: Muscle strength of the muscles in the thigh will be measured using an isokinetic dynamometer. Strength is measured by the amount of force (peak torque) and will be divided by body mass (kg). Strength is reported as a percent of body weight. A greater peak torque percentage is considered better.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percent body weight
Arm/Group | 4000 IU Vitamin D | 800 IU Vitamin D
Number analyzed (Participants) | 3 | 2
percent body weight | 58.9 (39.7) | 55.3 (16.7)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Subjects were under supervision for chronic kidney disease by physician
Arm/Group | 4000 IU Vitamin D | 800 IU Vitamin D
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT03710161/Prot_SAP_001.pdf